CLINICAL TRIAL: NCT02500342
Title: Effect of Thyroid Hormone Replacement on Fatigability in Untreated Older Adults With Subclinical Hypothyroidism
Acronym: TRUST FATIGUE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University College Cork (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 162/11_2
Record Dates: First submitted 2015-06-18; First posted 2015-07-16 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Thyroid Dysfunction; Mental Fatigue; Fatigue
Keywords: Thyroid Dysfunction; Fatigue; Randomized Controlled Trial; Thyroxine; Hypothyroidism
MeSH Terms: conditions — Mental Fatigue; Fatigue; Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: Levothyroxine (Experimental): The intervention will start with Levothyroxine 50 mcg daily (reduced to 25 mcg in subjects <50 kg of body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) vs. matching placebo; at 3 months, if the serum TSH level is <0.4 mU/L, dose will be reduced by 25 mcg; TSH >=0.4 and <4.6 mU/L, no change to dose; TSH >=4.6 mU/L, additional 25 mcg. The process will be repeated at 12 months, then annually; mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine which will be prescribed is 150 mcg (after 4 increments of 25 mcg at 3 months, 1, 2, 3 years; from the starting dose of 50 mcg).
  Interventions: Drug: Levothyroxine
- Drug: Placebo (Placebo Comparator): Control patients will obtain a placebo pill of the same characteristics as the intervention drug, and mock titration will be carried out identically to the intervention drug.
  Pharmaceutical composition of placebo (100 mg): Lactose monohydrate 66 mg, Maize starch 25 mg, Gelatin 5 mg, Croscarmellose sodium 3.5 mg, Magnesium stearate (vegetable source) 0.5 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxine — The intervention will start with Levothyroxine 50 mcg daily (reduced to 25 mcg in subjects <50 kg of body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) vs. matching placebo; at 3 months, if the serum TSH level is <0.4 mU/L, dose will be reduced by 25 mcg; TSH >=0.4 and <4.6 mU/L, no change to dose; TSH >=4.6 mU/L, additional 25 mcg. The process will be repeated at 12 months, then annually; mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine which will be prescribed is 150 mcg (after 4 increments of 25 mcg at 3 months, 1, 2, 3 years; from the starting dose of 50 mcg).
  Arms: Drug: Levothyroxine
Drug: Placebo — Control patients will obtain a placebo pill of the same characteristics as the intervention drug, and mock titration will be carried out identically to the intervention drug.
  Pharmaceutical composition of placebo (100 mg): Lactose monohydrate 66 mg, Maize starch 25 mg, Gelatin 5 mg, Croscarmellose sodium 3.5 mg, Magnesium stearate (vegetable source) 0.5 mg.
  Arms: Drug: Placebo

SUMMARY:
Thyroid hormone is a key regulatory hormone for a range of physiological systems. An impaired function of the thyroid gland such as subclinical hypothyroidism (SCH) can affect quality of life. Older adults with subclinical hypothyroidism often report non-specific symptoms such as tiredness. In addition, muscle symptoms such as cramps, weakness and myalgia are more common in SCH than in healthy controls. At present, evidence is lacking about the benefits of thyroxine replacement in the elderly with SCH, as no large randomized clinical trials (RCT) on the full range of relevant clinical outcomes, including tiredness have been performed. Moreover, there is continued uncertainty about the long-term impact on health related quality of life of thyroxine treatment for SCH. The aim of the study is to examine, within a large RCT of elderly participants with subclinical hypothyroidism, the impact of thyroxine therapy on the association between subclinical thyroid disease (SCTD) and the level of physical and mental fatigue. The existing trial infrastructure (TRUST thyroid trial-Euresearch FP7; clinicaltrials.gov ID: NCT 01660126) will be utilized to collect information on the level of physical and mental fatigue by using the Pittsburgh Fatigability Scale at baseline and at 1 year from 220 participants with persistent subclinical hypothyroidism randomized to either thyroxine or placebo.

DETAILED DESCRIPTION:
Background

Thyroid hormone is a key regulatory hormone for a range of physiological systems. An impaired function of the thyroid gland such as subclinical hypothyroidism (SCH) can affect quality of life. Older adults with subclinical hypothyroidism often report non-specific symptoms such as tiredness. In addition, muscle symptoms such as cramps, weakness and myalgia are more common in SCH than in healthy controls. At present, evidence is lacking about the benefits of thyroxine replacement in the elderly with SCH, as no large randomized clinical trials (RCT) on the full range of relevant clinical outcomes, including tiredness have been performed. Moreover, there is continued uncertainty about the long-term impact on health related quality of life of thyroxine treatment for SCH.

Objective

To examine, within a large RCT of elderly participants with subclinical hypothyroidism (the TRUST trial), the impact of thyroxine therapy on the association between subclinical thyroid disease (SCTD) and the level of physical and mental fatigue.

Methods

The existing trial infrastructure (TRUST thyroid trial-Euresearch FP7, clinicaltrials.gov ID: NCT 01660126) will be utilized to collect information on the level of physical and mental fatigue by using the Pittsburgh Fatigability Scale at baseline and at 1 year from 220 participants with persistent subclinical hypothyroidism randomized to either thyroxine or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling patients aged >= 65 years with subclinical hypothyroidism
* Written informed consent

Exclusion Criteria

* Subjects currently under Levothyroxine or antithyroid drugs (amiodarone, lithium)
* Recent thyroid surgery or radio-iodine (within 12 months)
* Grade IV NYHA heart failure
* Prior clinical diagnosis of dementia
* Recent hospitalization for major illness or elective surgery (within 4 weeks)
* Terminal illness
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects who are participating in ongoing RCTs of therapeutic interventions (including CTIMPs)
* Plan to move out of the region in which the trial is being conducted within the next 2 years (proposed minimum follow-up period)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 276 (Actual)
Dates: Start 2014-01; Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in level of physical and mental fatigue as assessed by the Pittsburgh Fatigability Scale (PFS) score | At 1 year of follow-up

SECONDARY OUTCOMES:
Level of physical and mental fatigue as assessed by the PFS score | At baseline and at 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, MD MAS, Principal Investigator — Clinic for General Internal Medicine, Bern University Hospital Bern
Locations (3):
- University College Cork, National University of Ireland, Cork, Ireland
- Switzerland (2):
  - Department of General Internal Medicine, Lausanne, Canton of Vaud
  - Clinic for General Internal Medicine, Bern University Hospital Bern, Bern

REFERENCES:
- [Background] Razvi S, Ingoe L, Keeka G, Oates C, McMillan C, Weaver JU. The beneficial effect of L-thyroxine on cardiovascular risk factors, endothelial function, and quality of life in subclinical hypothyroidism: randomized, crossover trial. J Clin Endocrinol Metab. 2007 May;92(5):1715-23. doi: 10.1210/jc.2006-1869. Epub 2007 Feb 13. PMID 17299073
- [Derived] Stuber MJ, Moutzouri E, Feller M, Del Giovane C, Bauer DC, Blum MR, Collet TH, Gussekloo J, Mooijaart SP, McCarthy VJC, Aujesky D, Westendorp R, Stott DJ, Glynn NW, Kearney PM, Rodondi N. Effect of Thyroid Hormone Therapy on Fatigability in Older Adults With Subclinical Hypothyroidism: A Nested Study Within a Randomized Placebo-Controlled Trial. J Gerontol A Biol Sci Med Sci. 2020 Sep 16;75(9):e89-e94. doi: 10.1093/gerona/glaa123. PMID 32577745